CLINICAL TRIAL: NCT05253755
Title: A Randomized, Observer-Blinded, Within Patient Bilateral Comparison to Study the Safety and Efficacy of Daily Application for 4 Weeks of DBI-001 Gel Versus Aqueous Gel in Subjects With Atopic Dermatitis
Brief Title: Study the Safety and Efficacy of DBI-001 Gel Versus Aqueous Gel
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor suspension and not due to safety or site-related matters.
Sponsor: DermBiont, Inc. (Industry)
Collaborators: Derm Research, PLLC (Other); Northsoundderm (Other); Clear Dermatology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DBI-207
Record Dates: First submitted 2021-11-01; First posted 2022-02-24 (Actual); Results first posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-10

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — BANG polymer gel

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DBI-001 Gel (Active Comparator): DBI-001 Gel: Topical application of DBI-001 gel on skin affected with atopic dermatitis.
  (This study is a within-subject bilateral controlled study)
  Interventions: Biological: DBI-001
- Aqueous Gel (Placebo Comparator): Aqueous Gel: Topical application of aqueous gel on skin affected with atopic dermatitis.
  (This study is a within-subject bilateral controlled study)
  Interventions: Biological: Aqueous gel

INTERVENTIONS:
Biological: DBI-001 — Topical application of DBI-001 gel on skin affected with atopic dermatitis.
  Arms: DBI-001 Gel
Biological: Aqueous gel — Topical application of aqueous gel on skin affected with atopic dermatitis.
  Arms: Aqueous Gel

SUMMARY:
The purpose for this study is to assess the Safety and Efficacy of Daily Application for 4 weeks of DBI-001 Gel Versus Aqueous Gel in Subjects with Atopic Dermatitis

DETAILED DESCRIPTION:
This is a randomized, observer blinded, Aqueous Gel-controlled, within-patient, bilateral comparison trial examining the effect of daily application for 4 weeks of DBI-001 Gel vs. Aqueous Gel on the clinical Atopic Dermatitis Severity Index (ADSI) scores and the abundance of Staphylococcus aureus of comparable bilateral target sites of Atopic Dermatitis (AD), as well as signs and symptoms of local tolerability on treated sites in subjects.

Subjects meeting the inclusion/exclusion criteria and having moderate to severe AD lesions at screening and baseline/Day 1 will be enrolled into the study.

In an observer-blinded fashion, each subject will have two sites randomly assigned to have either DBI-001 Gel or Aqueous Gel applied to the designated treatment targeted sites.

After Screening, Study visits will occur at Day 1 Baseline then Days 7 (±2), 14 (±2), 21 (±2), 28 (±2), 35 (±4), and 42 (±4)

ELIGIBILITY:
Inclusion Criteria:

* 1. Ability to understand, agree to, and sign the study Informed Consent. If the patient is unable to provide consent for him/herself, the patient's legally authorized representative may provide written consent.
* 2. A signed Health Information Portability and Accountability Act (HIPAA) authorization form which permits the use and disclosure of subject's individually identifiable health information.
* 3. Male or Female Subjects of any race 12 - 65 years of age.
* 4. Physician diagnosed clinically stable AD according to the criteria of Hanifin and Rajka with symmetrical bilateral target lesions (Hanifin and Rajka 1980). Lesion on each arm or leg must have an Atopic Dermatitis Severity Index (ADSI) ≥6. The 2 sites need to be comparable anatomically symmetrical sites. It will be in the opinion of the Investigator based on subject's medical history whether the lesions are clinically stable.
* 5. Female patients of child-bearing potential must use at least one method of birth control that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or vasectomized partner for the duration of study participation.
* 6. Technical ability and willingness to apply test articles during telemedicine visits with the study staff and unsupervised on weekends.
* 7. Willingness to discontinue use of systemic AD treatments and topical treatments to the target areas for the duration of the study unless specifically permitted by the Investigator.
* 8. Willingness to comply with test site restriction for 12 hours prior to all office visits including the Baseline visit and for 12 hours after each treatment application. These treatment site restrictions include:

  1. No washing of test sites with any cleansers or soaps at any time from the Baseline visit to completion of the Day 42 Follow up Visit. Water passing over the areas during showering is acceptable.
  2. No rubbing the test sites with a washcloth, towel, luffas. Pat dry after showering is acceptable.
  3. No recreational activities in chlorinated or chemically treated water such as swimming pools, hot tubs, and spas.
  4. No tight or form fitting clothing covering the treatment areas.
  5. No sunbathing or use of suntan parlors or tanning beds.
  6. If participating in physical activities resulting in heavy perspiration only pat dry test site areas with towel if needed.
  7. Any activity that in the opinion of the investigator might alter the quality of the samples collected or risk removal of the test article.
* 9. Willingness to undergo the following washout periods:

  1. Washout of 2 weeks prior to the Baseline visit for topical treatments used on the two treatment target sites, including but not limited to: antibacterial products, anti-inflammatories (e.g., corticosteroids, tacrolimus, Pimecrolimus). Other than the two sites on the arms or legs, topical medications may be used before/during the duration of the study. Subjects will be provided 1% hydrocortisone for treating non-target areas during the trial.
  2. Washout of 4 weeks prior to the Baseline visit for systemic treatments for AD, including but not limited to corticosteroids (oral or intramuscular injections), systemic immunomodulators or immunosuppressive (e.g., methotrexate, cyclosporine, hydroxychloroquine), antibiotics (oral or injected, if required to treat a medical condition short duration of oral antibiotics (≤10 days) are permitted after randomization)
  3. Washout of 2 weeks prior to the Baseline visit for bleach baths.
  4. Washout of 2 weeks prior to the Baseline visit for phototherapy.
* 10. No history of allergy to at least two of the following classes of antibiotics: Cephalosporin, Quinolone, Tetracycline, Aminoglycosides Macrolide, Carbapenems and Lipopeptides.
* 11. Willingness to allow digital photos of arms or legs to be taken and stored.

Exclusion Criteria:

* 1. Women who are pregnant, planning a pregnancy, breastfeeding or have a positive pregnancy test at screening.
* 2. Any dermatological conditions that could interfere with clinical evaluations or any disease state or physical condition which might expose the patient to an unacceptable risk by study participation.
* 3. Any underlying disease(s) or other dermatological conditions that require the use of exclusionary topical or systemic therapy.
* 4. Spontaneously improving or rapidly deteriorating dermatitis anywhere on the body.
* 5. Netherton's syndrome or other genetic dermatoses that result in defective epidermal barrier function.
* 6. Treatment of any type of cancer within the last 6 months other than cutaneous basal cell carcinoma.
* 7. History of any significant internal disease (which contraindicates use of live microbiome e.g. leukemia, liver failure, cardiovascular disease).
* 8. Subjects who are known to be allergic to any of the test product(s) or any components in the test product(s) or history of hypersensitivity or allergic reactions to any of the study preparations as described in the Investigator's Brochure.
* 9. AIDS or AIDS related complex by medical history.
* 10. Known or suspected immune suppressive medications or diseases or any condition that in the opinion of the investigator would increase the subject's susceptibility to opportunistic infections. 11. Treatment with systemic immune modulating or anti-inflammatory biologics agents within 16 weeks of Baseline Visit.
* 12. Poorly controlled diabetes mellitus Type I or II by medical history.
* 13. Peripheral vascular disease based on medical history.
* 14. Any subject not able to meet the study attendance and telemedicine visit requirements.
* 15. Participants with a history of psychiatric disease or history of alcohol or drug abuse that would interfere with the ability to comply with the study protocol.
* 16. Subjects who have participated in any other trial of an investigational drug or device within 30 days prior to enrollment or participation in a research study concurrent with this study.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Investigate MD, LLC, Scottsdale, Arizona
  - DermResearch, Inc., Austin, Texas
  - North Sound Dermatology, Mill Creek, Washington

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: bilateral target lesions
Groups:
- DBI-001 Gel and Aqueous Gel: DBI-001: Topical application of DBI-001 gel on skin affected with atopic dermatitis.
  Aqueous Gel: Topical application of aqueous gel on skin affected with atopic dermatitis.
Period: Overall Study
Arm/Group | DBI-001 Gel and Aqueous Gel
Started | 10; 20 bilateral target lesions
Completed | 9; 18 bilateral target lesions
Not Completed | 1; 2 bilateral target lesions

BASELINE CHARACTERISTICS:
Groups:
- DBI-001 and Aqueous Gel: DBI-001: Topical application of DBI-001 gel on skin affected with atopic dermatitis.
  Aqueous gel: Topical application of aqueous gel on skin affected with atopic dermatitis.
  (This study is a within-subject bilateral controlled study)
Arm/Group | DBI-001 and Aqueous Gel
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] — Subjects were 12 to 65 years old with a mean age of 30.8 years. The majority of participants were female(60%).
  years | 30.8 (14.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Individual Signs and Symptoms of Atopic Dermatitis
Description: Change from baseline in individual signs and symptoms of Atopic Dermatitis (components of the ADSI score) at days 7, 14, 21, 28, 35, and 42 of sites treated with DBI-001 Gel or Aqueous Gel Atopic Dermatitis Severity Index: The ADSI score represents the sum of the individual severity scores of none, mild, moderate, or severe for the following component signs and symptoms: erythema, pruritus, exudation, excoriation, and lichenification. To calculate the ADSI score, the component scores are added together.
  Scale for the individual components:
  0=none
  1. mild
  2. moderate
  3. severe
Time Frame: 42 days of participation
Population: This study is a within-subject bilateral controlled study.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- DBI-001 Gel: Topical application of DBI-001 gel on skin affected with atopic dermatitis.
Arm/Group | DBI-001 Gel | Aqueous Gel
Number analyzed (Participants) | 8 | 8
score on a scale
  Erythema Day 0 | 2 [2 to 2] | 2 [2 to 2]
  Erythema Day 7 | 2 [2 to 2] | 2 [1.75 to 2]
  Erythema Day 14 | 2 [1 to 2] | 1.5 [1 to 2]
  Erythema Day 21 | 2 [1 to 2] | 1.5 [1 to 2]
  Erythema Day 28 | 1 [1 to 1.25] | 1 [0.75 to 1.25]
  Erythema Day 35 | 1 [1 to 2] | 1.5 [1 to 2]
  Erythema Day 42 | 1.5 [1 to 2] | 1 [1 to 2]
  Pruritus Day 0 | 2 [1.75 to 2] | 2 [1 to 2]
  Pruritus Day 7 | 1.5 [1 to 2] | 1.5 [1 to 2.25]
  Pruritus Day 14 | 1 [1 to 1.25] | 1 [1 to 2]
  Pruritus Day 21 | 1 [0 to 1] | 1 [0.75 to 2]
  Pruritus Day 28 | 1 [0 to 1] | 1 [0.75 to 2]
  Pruritus Day 35 | 1 [0.75 to 1.25] | 1.5 [0.75 to 2]
  Pruritus Day 42 | 1 [0 to 1.25] | 1 [0 to 2]
  Exudation Day 0 | 0.5 [0 to 1] | 0.5 [0 to 1]
  Exudation day 7 | 1 [0.75 to 1] | 0.5 [0 to 1]
  Exudation day 14 | 0.5 [0 to 1] | 0 [0 to 1]
  Exudation day 21 | 0.5 [0 to 1] | 0 [0 to 1]
  Exudation day 28 | 0.5 [0 to 1] | 0 [0 to 1]
  Exudation day 35 | 0.5 [0 to 1] | 0 [0 to 1]
  Exudation day 42 | 0 [0 to 1] | 0 [0 to 0]
  Excoriation Day 0 | 1 [1 to 2] | 1 [1 to 2]
  Excoriation Day 7 | 1 [1 to 1.25] | 1 [1 to 1]
  Excoriation Day 14 | 1 [0 to 1.25] | 1 [0 to 1]
  Excoriation Day 21 | 1 [0 to 1.25] | 1 [0 to 1.25]
  Excoriation Day 28 | 1 [0 to 2] | 0.5 [0 to 1.25]
  Excoriation Day 35 | 1 [0 to 1] | 1 [0 to 1]
  Excoriation Day 42 | 1 [0.75 to 1] | 1 [0 to 1]
  Lichenification Day 0 | 2 [1 to 2] | 2 [1.75 to 2]
  Lichenification Day 7 | 2 [1 to 2] | 2 [1.75 to 2]
  Lichenification Day 14 | 2 [1 to 2] | 2 [1 to 2]
  Lichenification Day 21 | 2 [1.75 to 2] | 2 [1.75 to 2]
  Lichenification Day 28 | 2 [1 to 2] | 2 [1 to 2]
  Lichenification Day 35 | 2 [1 to 2] | 2 [1 to 2]
  Lichenification Day 42 | 2 [1 to 2] | 2 [1 to 2]

ADVERSE EVENTS:
Time Frame: Approximately 56 days. Timeframe details of the 4 adverse events: Pruritus started after Baseline visit and resolved before Day 7 Emesis started after Day 7 and resolved before Day 14 Erythematous papules started after Day 28 visit and resolved before Day 35 visit Gout Flare started on Day 14
Arm/Group | DBI-001 Gel | Aqueous Gel
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 2/10 | 2/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DBI-001 Gel (N=10) | Aqueous Gel (N=10)
Emesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Allergic Reaction to cats (pruritus) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythematous papules (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Gout flare (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT05253755/Prot_SAP_000.pdf